CLINICAL TRIAL: NCT03609879
Title: Effect of Cervical Collar on Optic Nerve Sheath Diameter Measured Sonographically. A Randomized Crossover Trial
Brief Title: Effect of Cervical Collar on Intracranial Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazarski University (Other)
Collaborators: Wroclaw Medical University (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Associate Professor, Lazarski University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ONSD_2018_UL
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Optic Nerve Sheath Diameter; Ultrasonography
Keywords: cervical collar; sonography; adult patients; Optic nerve sheath diameter; Ultrasonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without cervical collar (No Intervention): baseline - without cervical collar
- with cervical collar (Experimental): scenarios with cervical collars
  Interventions: Device: Ambu Perfect ACE; Device: Philly One-Peace Collar; Device: Necloc Collar; Device: NexSplit Plus; Device: NECKLITE

INTERVENTIONS:
Device: Ambu Perfect ACE — patient with a fitted cervical collar (Ambu Perfect ACE) established by an experienced instructor. Cervical collar set up for 20 minutes
  Arms: with cervical collar
Device: Philly One-Peace Collar — patient with a fitted cervical collar (Philly One-Peace Collar) established by an experienced instructor. Cervical collar set up for 20 minutes
  Arms: with cervical collar
Device: Necloc Collar — patient with a fitted cervical collar (Neclock Collar) established by an experienced instructor. Cervical collar set up for 20 minutes
  Arms: with cervical collar
Device: NexSplit Plus — patient with a fitted cervical collar (NexSplit Plus) established by an experienced instructor. Cervical collar set up for 20 minutes
  Arms: with cervical collar
Device: NECKLITE — patient with a fitted cervical collar (NECKLITE) established by an experienced instructor. Cervical collar set up for 20 minutes
  Arms: with cervical collar

SUMMARY:
The routine use of cervical collar in emergency medical conditions has recently been questioned. The application of cervical collars, as their opponents point out, results in deterioration of intubation conditions, intensification of pain in the region of mastoid processes, and impaired venous outflow from the head.

ELIGIBILITY:
Inclusion Criteria:

* voluntary participation in the study

Exclusion Criteria:

* head or the spine injury in the last 3 months
* eye injuries in the last 3 months
* amputation of the eyeball
* Headache

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter 5 minutes after collar placement | 1 day after
  During each evaluation with Optic nerve sheath diameter, at least three measurements were attempted from each eye. The ONSD was measured 3 mm behind the retina. All scans were performed using a 13-6 MHz linear-array probe and a high resolution optimization setting.
Optic nerve sheath diameter 20 minutes after collar placement | 1 day after
  During each evaluation with Optic nerve sheath diameter, at least three measurements were attempted from each eye. The ONSD was measured 3 mm behind the retina. All scans were performed using a 13-6 MHz linear-array probe and a high resolution optimization setting.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Lazarski University
Locations (2):
- Poland (2):
  - Faculty of Medicine, Lazarski University, Warsaw, Masovian Voivodeship
  - Lazarsku University, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided
Research data will be available from the principal investigator

REFERENCES:
- [Background] Szarpak L, Truszewski Z, Kurowski A, Samarin S, Evrin T, Adamczyk P, Czyzewski L. Knowledge, attitude, and practices of paramedics regarding optic nerve sheath diameter ultrasonography. Am J Emerg Med. 2016 Jun;34(6):1160-1. doi: 10.1016/j.ajem.2016.02.063. Epub 2016 Mar 3. No abstract available. PMID 26994678
- [Derived] Ladny M, Smereka J, Ahuja S, Szarpak L, Ruetzler K, Ladny JR. Effect of 5 different cervical collars on optic nerve sheath diameter: A randomized crossover trial. Medicine (Baltimore). 2020 Apr;99(16):e19740. doi: 10.1097/MD.0000000000019740. PMID 32311968